CLINICAL TRIAL: NCT03532035
Title: A Randomized, Controlled, Open-Label, Multiple Ascending Dose Study of Intravenous Brincidofovir in Adult Allogeneic Hematopoietic Cell Transplant Recipients With Adenovirus Viremia
Brief Title: Open Label Study of IV Brincidofovir in Adult Transplant Recipients With Adenovirus Viremia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: terminated due to low enrollment rate
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMX001-211
Record Dates: First submitted 2018-04-26; First posted 2018-05-22 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Adenovirus
MeSH Terms: conditions — Adenoviridae Infections | interventions — brincidofovir; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brincidofovir (BCV) (Experimental): * Cohort 1: BCV 10 mg twice weekly via IV infusion over 2 hours
  * Cohort 2: BCV 15 mg twice weekly via IV infusion over 2 hours
  * Cohort 3: BCV In Cohort 3, the actual dose may be higher or lower than doses administered in previous cohorts; the maximum dose of IV BCV will be ≤ 25 mg.
  Interventions: Drug: Brincidofovir
- Standard of Care (SoC) (Active Comparator): Subjects randomized to the SoC in each cohort will be managed per local institutional guidelines and investigator judgement. SoC treatment options may include, but are not limited to, taking a "watch and-wait" approach, with or without decreased immunosuppression (i.e., no active treatment), or treatment with IV Cidofovir (CDV), ganciclovir, or ribavirin.
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Brincidofovir — Subjects will receive BCV administered as a continuous IV infusion over 2 hours twice weekly (on Days 1, 4, 8, and 11) for a period of 2 weeks (total of 4 doses).
  Other Names: BCV
  Arms: Brincidofovir (BCV)
Drug: Standard of Care — Subjects randomized to the SoC in each cohort will be managed per local institutional guidelines and investigator judgement. SoC treatment options may include, but are not limited to, taking a "watch and-wait" approach, with or without decreased immunosuppression (i.e., no active treatment), or treatment with IV CDV, ganciclovir, or ribavirin.
  Arms: Standard of Care (SoC)

SUMMARY:
This is a randomized, controlled, open-label, multicenter study to evaluate the safety, tolerability, pharmacokinetic (PK), and adenovirus (AdV) antiviral activity of multiple ascending doses of IV brincidofovir (BCV). Approximately 30 eligible subjects will be sequentially enrolled into 1 of 3 planned cohorts. Within each cohort, subjects will be randomized in a 4:1 ratio to receive IV BCV dosed twice weekly (BIW) (on Days 1, 4, 8, and 11) or to receive investigator-assigned standard of care (SoC).

ELIGIBILITY:
Inclusion Criteria:

* Be ≥ 18-years-old (or per local law or regulations on legal age of consent).
* Have received an allogeneic hematopoietic cell transplant (HCT) within the previous 100 days.
* Have plasma AdV DNA viremia ≥ 1,000 copies/mL (via quantitative polymerase chain reaction assay; local results must be confirmed by the designated central virology laboratory).

Exclusion Criteria:

* Diarrhea meeting the US National Institutes of Health (NIH)/National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 or greater
* Acute graft versus host disease (GVHD)

  1. NIH Stage 2 or higher acute GVHD of the gut (i.e., diarrhea > 1,000 mL/day, or severe abdominal pain with or without ileus) or liver (i.e., bilirubin > 3 mg/dL : > 51 μmol/L) within 7 days prior to Day 1
  2. Any NIH Stage 3 or Stage 4 acute GVHD within 7 days prior to Day 1
* Concurrent human immunodeficiency virus or active hepatitis B or C infection
* An estimated creatinine clearance of < 30 mL/min, and/or use of renal replacement therapy within 7 days prior to Day 1.
* Poor clinical prognosis, including active malignancy, irreversible organ failure, use of vasopressors, requirement for mechanical ventilation, resting oxygen saturation < 88%, or Pulmonary Arterial oxygen (PaO2) ≤ 55 mm Hg without supplemental oxygen at any time within 7 days prior to Day 1.
* Receiving or anticipated to start systemic cyclosporine immunosuppressant treatment during study participation.
* Received treatment with CDV within 14 days prior to Day 1.
* Previous receipt of cell-based anti-AdV therapy within 6 weeks prior to Day 1 or prior receipt of an anti-AdV vaccine at any time.
* Consumed food products containing sesame seeds, sesame oil, or dietary supplements containing sesamin within 3 days prior to Day 1.
* Received any investigational drug within 28 days prior to Day 1 or currently participating in another interventional study.
* Pregnant or breastfeeding.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Plasma area under the curve (AUC) of BCV | 15 days
  BCV AUC will be determined by analysis of BCV plasma concentrations at the following time points after the start of Dose 1 and Dose 4: 30 minutes, and 2.5, 3, 4, 8, 10, 12, 36, and 72 hours
Plasma Cmax of BCV | 15 days
  BCV Cmax will be determined by analysis of BCV plasma concentrations at the following time points after the start of Dose 1 and Dose 4: 30 minutes, and 2.5, 3, 4, 8, 10, 12, 36, and 72 hours
Incidence (number and percentage of subjects) of treatment-emergent adverse events | 22 days

CONTACTS AND LOCATIONS:
Locations (8):
- United States (4):
  - UCLA Medical Center, Los Angeles, California
  - University of Chigago, Chicago, Illinois
  - Brigham and Womens Hospital, Boston, Massachusetts
  - MD Anderson Cancer Center, Houston, Texas
- University Vita-Salute San Raffaele. San Faffaele Scientific Institute, Milan, Italy
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitari I Politecnic la Fe, Valencia